CLINICAL TRIAL: NCT06447727
Title: Efficacy and Safety of 90Y Microsphere Combined With FOLFIRI and Bevacizumab in Second-line Treatment of Colorectal Cancer Liver Metastasis
Brief Title: Efficacy and Safety of 90Y Microsphere Combined With FOLFIRI and Bevacizumab in Second-line Treatment of CRLM
Status: Recruiting | Type: Observational
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Gao-jun Teng, Dean, Zhongda Hospital
Other Study IDs: ST-Y90-CP01
Record Dates: First submitted 2024-06-03; First posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Colorectal Cancer Metastatic
Keywords: Yttrium[90Y]; colorectal cancer liver metastases, CRLM
MeSH Terms: interventions — Sirtuins; Bevacizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SIRT with Yttrium-90 Microspheres combined with FOLFIRI and Bevacizumab: Selective Internal Radiation Therapy (SIRT) with Yttrium-90 [90Y] Microspheres Injection combined with FOLFIRI and Bevacizumab
  Interventions: Drug: SIRT with Yttrium-90 Microspheres; Drug: FOLFIRI and Bevacizumab

INTERVENTIONS:
Drug: SIRT with Yttrium-90 Microspheres — Selective Internal Radiation Therapy (SIRT) with Yttrium-90 [90Y] Microspheres Injection
Drug: FOLFIRI and Bevacizumab — FOLFIRI and Bevacizumab

SUMMARY:
To observe the PFS of yttrium [90Y] microsphere injection combined with FOLFIRI and bevacizumab in second-line treatment of CRLM.

DETAILED DESCRIPTION:
This study is a prospective, multicenter, observational, cohort study to observe the efficacy and safety of selective internal radiation therapy (SIRT) with yttrium [90Y] microsphere injection combined with FOLFIRI and bevacizumab as second-line therapy in patients with colorectal cancer liver metastases.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old≤ age ≤ 75 years old
2. Voluntarily signed informed consent
3. Patients with liver metastases of colorectal cancer, colorectal cancer lesions have resection, liver metastases limited to a single lobe
4. The liver tumor progresses after first-line treatment, and FOLFIRI combined with bevacizumab therapy is planned
5. On the assessment of the clinician, the patient was eligible for yttrium [90Y] microspheres injection, and treatment with yttrium [90Y] microspheres injection was planned
6. KRAS mutant
7. ECOG PS: 0-1
8. Child Pugh score ≤7
9. Adequate level of organ function：a) Hematology: Neutrophils (ANC) ≥1.5×109/L, hemoglobin (HB) ≥90 g/L, platelets (PLT) ≥75×109/L；b) Liver function: albumin > 3 g/dL; ALT and AST≤ 5 x ULN; TBIL < 34.0 μmol/L；c) Renal function: serum creatinine ≤176.8 μmol/L or endogenous creatinine clearance > 50 mL/min；d) Coagulation function: INR≤1.2.

Exclusion Criteria:

1. After liver metastasis was diagnosed, the liver underwent external radiation therapy and transhepatic arterial chemoembolization
2. Patients with extrahepatic metastases
3. Pregnant and lactating women
4. History of severe arrhythmia or heart failure
5. Other researchers considered it inappropriate to participate in this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with liver metastasis of colorectal cancer
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival(PFS) | until death or 18 months after treatment with yttrium [90Y] microspheres, whichever occurred first.
  Defined as the time from the start of FOLFIRI treatment to the date of radiographic progression or death due to any cause, whichever occurs first, based on RECIST 1.1 criteria.

SECONDARY OUTCOMES:
Objective response rate（ORR） | until death or 18 months after treatment with yttrium [90Y] microspheres, whichever occurred first.
  defined as the time between the date of initiation of treatment with FOLFIRI and the date of radiographic progression or death from any cause, whichever occurs first. According to RECIST 1.1 criteria.
Disease control rate (DCR) for target lesions | until death or 18 months after treatment with yttrium [90Y] microspheres, whichever occurred first.
  defined as the proportion of subjects who achieve optimal tumor response or stable disease (complete response, partial response, or stable disease) over the course of the study. Assessed according to RECIST 1.1 criteria.
Conversion resection rate | until death or 18 months after treatment with yttrium [90Y] microspheres, whichever occurred first.
  the proportion of participants who underwent successful surgical resection of unresectable CRLM after receiving SIRT in combination with FOLFIRI and bevacizumab.
Hepatic progression-free survival (hPFS) | until death or 18 months after treatment with yttrium [90Y] microspheres, whichever occurred first.
  defined as the time between the date of initiation of treatment with FOLFIRI and the date of progression on liver imaging or death from any cause, whichever occurs first. Assessed according to RECIST 1.1 criteria.
Overall survival (OS) | until death or 18 months after treatment with yttrium [90Y] microspheres, whichever occurred first.
  defined as the time between the date of initiation of treatment with FOLFIRI and the date of death due to any cause.
Safety(adverse events) | within 6 months from the start of SIRT treatment.
  Incidence of grade 3 and above adverse events (NCI-CTCAE v5.0) within 6 months from the start of SIRT treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Gao-Jun Teng, Principal Investigator — Zhongda Hospital
Locations (1):
- Zhongda Hospital，Southeast University, Nanjing, Jiangsu, China